CLINICAL TRIAL: NCT06132854
Title: Efficacy of Virtual Reality Based Simulation in the Preparation of Children for Magnetic Resonance Imaging Examinations: a Randomized Clinical Trial (MRVR)
Brief Title: VR Based Simulation in the Preparation of Children for MRI - MRVR
Acronym: MRVR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Semmelweis University (Other)
Responsible Party: Principal Investigator, Dr. Horváth Klára, assistant professor, Semmelweis University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: SE RKEB 202/2021
Record Dates: First submitted 2023-11-06; First posted 2023-11-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Children, Only; Anesthesia
Keywords: MRI; Pediatrics; anesthesia; virtual reality

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants cannot be blinded due to the nature of the study. The radiologists, anesthesiology team, MRI staff and the second research assistant administering post-procedure questionnaires and coding anesthesiology data intended to be blinded, however, children may disclose their group by talking about their experience.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- VR (Experimental): Participants in the VR group are immersed in a unique 360° VR experience specifically designed for this study.
  The custom made VR experience consists of two parts. In the first part, children find themselves in a simulated MRI room which resembles to the one they will be scanned.
  The second half of the VR experience introduces a mindfulness-ACT based meditation segment within the context of a space travel.
  Interventions: Other: VR
- Booklet (Active Comparator): Children in the booklet condition will be prepared by using an educational booklet containing colorful illustrations of the MRI examination room and about the procedure. This serves as a resource to familiarize them with the MRI procedure, address common concerns, and provide information about what to expect during the exam. The role of the booklet condition is to serve as an active control for our experimental condition. This condition also contains an interaction with the experimenter and increases familiarity through explanation and illustrations. However, it does not involve the immersive effect of the VR.
  Interventions: Other: Booklet
- Usual care (No Intervention): In the usual care condition children are prepared by the healthcare staff through explanations, reframing, playing as per personal preference which is currently the standard of care in our departments.

INTERVENTIONS:
Other: VR — The virtual environment is provided by the Oculus Quest 2 or 3 VR headset, providing a high-quality and immersive visual experience.
  Arms: VR
Other: Booklet — Children in the booklet condition will be prepared by using an educational booklet containing colorful illustrations of the MRI examination room and about the procedure.
  Arms: Booklet

SUMMARY:
The goal of this randomized controlled trial is to evaluate whether a virtual reality based preparation method can efficiently decrease the proportion of children requiring general anesthesia during MRI examinations.

Participants will take part in a virtual reality environment resembling an MRI before their scheduled MRI examination.

Researchers will compare these children to usual care and a booklet based preparation method to see if less children need anesthesia for completing the MRI examination.

DETAILED DESCRIPTION:
Study Description:

Our study investigates the efficacy of a custom-made virtual reality experience in the preparation of children for MRI examinations. We hypothesise that preparation with VR can significantly reduce the need for anesthesia in children during MRI examinations, or if anesthesia is needed less doses of anesthetics are required.

Objectives:

Primary Objective:

To evaluate whether the VR based preparation decreases the need for anesthesia and sedation during MRI examinations.

Secondary Objectives:

To evaluate whether fear, mood, anxiety, familiarity with the MRI examination of the children and willingness to take part again change as a result of the intervention.

Endpoints:

Primary Endpoint:

The need for any anesthetic or sedative medication during MRI examination.

Secondary Endpoints:

Visual analogue scales related to fear, mood and familiarity, willingness to take part in an MRI examination again.

Study Population: 288 children aged 4-18 years who are in- or outpatients at the Pediatric Center of the Semmelweis University and are scheduled for MRI examination with anesthesia will be enrolled.

Description of Sites/Facilities Enrolling Participants:

The study takes place in the two Departments of the Pediatric Centre of the Semmelweis University

Description of Study Intervention/Experimental Manipulation:

Our research will be conducted as a three arm randomized controlled trial (VR, booklet, usual care). Participants in the VR condition are immersed in a unique 360° VR experience specifically designed for this study.

Children in the booklet condition will be prepared by using an educational booklet containing colorful illustrations about the MRI examination.

In the usual care condition children are prepared by the healthcare staff without using any specific equipment or standardized methods.

Study Duration:

36 months

Participant Duration:

All participants need a single visit intervention to complete all study related tasks.

ELIGIBILITY:
Inclusion Criteria:

1. Informed assent and parental informed consent to participate in the study.
2. Stated willingness to participate in the intervention and to complete study questionnaires.
3. Inpatient or outpatient at the Pediatric Center.
4. Age 4-18 years
5. Scheduled for MRI examination under anesthesia at the Semmelweis University.
6. Fluent in Hungarian language

Exclusion Criteria:

1. Severe visual impairment or hearing loss that would hinder the participation of the VR and booklet experience.
2. In case of epilepsy, if the treating physician recommend against participation.
3. Children with severe intellectual disability which would hinder participation in the VR group e.g. not able to follow simple instructions.
4. Inpatients, if the treating physician indicates that the child is too unwell for the study.
5. Face or cranial deformities, wounds on the face and head which would hinder wearing the VR headset.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 288 (Estimated)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
proportion of children requiring anesthesia | during the MRI examination, assessed directly after the MRI from anesthesiology documentation
  proportion of children requiring any form of anesthesia or sedation during the MRI examination

SECONDARY OUTCOMES:
fear | assessed directly before the intervention, directly before the MRI examination, no later than 4 hours after the MRI examination
  fear of the child measured on a visual analogue scale range 1-100, higher indicating increased fear
mood | directly before the intervention, directly before the MRI examination, no later than 4 hours after the MRI examination
  mood of the child measured on a visual analogue scale, scale range 1-100, higher indicating better mood
nervousness | directly before the intervention, directly before the MRI examination, no later than 4 hours after the MRI examination
  nervousness of the child measured on a visual analogue scale, scale range 1-100, higher increased nervousness
familiarity | directly before the intervention, directly before the MRI examination, no later than 4 hours after the MRI examination
  familiarity of the child with the MRI examination measured on a visual analogue scale scale range 1-100, higher indicating increased familiarity with the MRI
willingness to take part again | no later than 4 hours after the MRI examination
  willingness of the child to take part in a future MRI examination measured on a visual analogue scale, scale range 1-100, higher indicating more willingness taking part in a future MRI examination
helpfulness | directly before the MRI examination
  indication how much the child found the preparation method helpful, measured on a visual analogue scale, scale range 1-100, higher indicating the preparation method was more helpful

OTHER OUTCOMES:
fear of the parent | directly before the intervention, directly before the MRI examination, no later than 4 hours after the MRI examination
  fear of the parent measured on a visual analogue scale, range 1-100, higher indicating increased fear
mood of the parent | directly before the intervention, directly before the MRI examination, no later than 4 hours after the MRI examination
  mood of the parent measured on a visual analogue scale, scale range 1-100, higher indicating better mood
nervousness of the parent | directly before the intervention, directly before the MRI examination, no later than 4 hours after the MRI examination
  nervousness of the parent measured on a visual analogue scale, scale range 1-100, higher increased nervousness
familiarity of the parent | directly before the intervention, directly before the MRI examination, no later than 4 hours after the MRI examination
  familiarity of the parent with the MRI examination measured on a visual analogue scale, scale range 1-100, higher indicating increased familiarity with the MRI
fear of the child assessed by parent | directly before the intervention, directly before the MRI examination, no later than 4 hours after the MRI examination
  fear of the child assessed by parent measured on a visual analogue scale, range 1-100, higher indicating increased fear
mood of the child assessed by parent | directly before the intervention, directly before the MRI examination, no later than 4 hours after the MRI examination
  mood of the child assessed by parent measured on a visual analogue scale, scale range 1-100, higher indicating better mood
nervousness of the child assessed by parent | directly before the intervention, directly before the MRI examination, no later than 4 hours after the MRI examination
  nervousness of the child assessed by parent measured on a visual analogue scale, scale range 1-100, higher increased nervousness
familiarity of the child assessed by parent | directly before the intervention, directly before the MRI examination, no later than 4 hours after the MRI examination
  familiarity of the child with the MRI examination assessed by parent measured on a visual analogue scale, scale range 1-100, higher indicating increased familiarity with the MRI
propofol dose | during the MRI examination, assessed from anesthesiology documentation 1 day after the MRI at the latest
  Dose of propofol used per body weight and duration of MRI examination.

CONTACTS AND LOCATIONS:
Overall Officials: Klara Horvath, MD PhD, Principal Investigator — Semmelweis University
Locations (1):
- Pediatric Center, Semmelweis University, Budapest, Budapest, Hungary

IPD SHARING:
Plan to Share IPD: No